CLINICAL TRIAL: NCT00252525
Title: CSP #465B - Correlation of Plasma Endothelial Cell (Basic Fibroblast Growth Factor) Activity With Cardiovascular Events In Patients With Diabetes Mellitus Type 2
Brief Title: Correlation of Plasma Endothelial Cell Activity With Cardiovascular Events in Patients With Diabetes Mellitus Type 2
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 465B
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: None Retained — The cohort consisted of patients that participated in the 465 main study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: This is an observational study of patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2@.

SUMMARY:
CSP 465-B, Correlation of Plasma Endothelial Cell (Basic Fibroblast Growth Factor) Activity With Cardiovascular Events in Patients with Diabetes Mellitus, Type II.

Mark Zimering M.D.

Objectives: Endothelial cell dysfunction plays a role in the development of the atherosclerotic vascular lesion and it is also thought to provide a mechanism for increased urinary albumin excretion in type 2 diabetes mellitus. Micro- or macroalbuminuria are associated with increased cardiovascular (CV) morbidity and mortality in type 2 diabetes mellitus. In at least one longitudinal study in older-age onset patients, micro-or macroalbuminuria robustly predicted increased CV risk independent of other diabetes-related factors.1 The pathogenetic mechanisms underlying a significant association between micro- or macroalbuminuria and CV risk in diabetes mellitus are not known but may include: growth factors, clotting factors, lipids, or hemodynamic factors. The aim of the present study is to investigate whether an angiogenic growth factor, basic fibroblast growth factor (bFGF), plays a role in increased CV risk in type 2 diabetes mellitus. Research Plan: BFGF (FGF-2) is one of the most potent known angiogenesis factors. Increased bFGF was previously associated with both endothelial cell injury and micro- or macroalbuminuria. In a prior study of 73 older-age onset veterans with type 2 diabetes mellitus (JCEM, 1996), we found plasma endothelial cell (bFGF) activity was significantly associated with glycemic levels, and (in multiple regression analysis) independently associated with both microalbuminuria and retinopathy. We will test whether plasma endothelial cell (bFGF) activity is significantly, independently associated with a pooled endpoint of cardiovascular events that includes myocardial infarction (MI), coronary revascularization, congestive heart failure (CHF), or CV mortality. We expect that increased bFGF may itself be a robust marker for increased CV risk in diabetes mellitus for three reasons. First, because bFGF was independently associated with (micro)-albuminuria in type 2 diabetes mellitus. Second, because increased bFGF was associated with increased activity in the renin-angiotensin system in vascular smooth muscle cells (Dzau, et al. JCI, 1995). And third, because (as we reported) angiotensin converting enzyme inhibitor (ACEi) drugs substantially decreased plasma bFGF levels in (micro)- albuminuric diabetes mellitus type 2, and (as others reported) ACEi drugs substantially reduced the risk of development of CHF in patients with LVH 2, the risk of mortality after MI (8,9), and the risk of CV death in diabetic patients with proteinuria.

Because plasma endothelial cell (bFGF) activity correlated significantly with glycemic levels in diabetes mellitus type 2, plasma bFGF may be one of the pathogenetic links between glycemic levels and an increased risk of cardiovascular events in diabetes mellitus, type 2.

Methods: Blood (3 mL EDTA plasma) will be collected from each subject in Years 1, and 2 of the Study at each of 6 local participating VA substudy sites. Because plasma endothelial cell (bFGF-like) bioactivity and bFGFR-IR in vivo are stable for months and years based on our prior published studies (1-3), we anticipate that obtaining 2 specimens, 1 each in Years 1, 2 of the study, will provide sufficient data to model proportional risk.

DETAILED DESCRIPTION:
Primary Hypothesis: The aim of the present study is to investigate whether an angiogenic growth factor, basic fibroblast growth factor (bFGF), plays a role in increased CV risk in type 2 diabetes mellitus.

Secondary Hypotheses:

Primary Outcomes: cardiovascular morbidity and mortality

Study Abstract:

CSP 465-B, Correlation of Plasma Endothelial Cell (Basic Fibroblast Growth Factor) Activity With Cardiovascular Events in Patients with Diabetes Mellitus, Type II.

Mark Zimering M.D.

Objectives: Endothelial cell dysfunction plays a role in the development of the atherosclerotic vascular lesion and it is also thought to provide a mechanism for increased urinary albumin excretion in type 2 diabetes mellitus. Micro- or macroalbuminuria are associated with increased cardiovascular (CV) morbidity and mortality in type 2 diabetes mellitus. In at least one longitudinal study in older-age onset patients, micro-or macroalbuminuria robustly predicted increased CV risk independent of other diabetes-related factors.1 The pathogenetic mechanisms underlying a significant association between micro- or macroalbuminuria and CV risk in diabetes mellitus are not known but may include: growth factors, clotting factors, lipids, or hemodynamic factors. The aim of the present study is to investigate whether an angiogenic growth factor, basic fibroblast growth factor (bFGF), plays a role in increased CV risk in type 2 diabetes mellitus. Research Plan: BFGF (FGF-2) is one of the most potent known angiogenesis factors. Increased bFGF was previously associated with both endothelial cell injury and micro- or macroalbuminuria. In a prior study of 73 older-age onset veterans with type 2 diabetes mellitus (JCEM, 1996), we found plasma endothelial cell (bFGF) activity was significantly associated with glycemic levels, and (in multiple regression analysis) independently associated with both microalbuminuria and retinopathy. We will test whether plasma endothelial cell (bFGF) activity is significantly, independently associated with a pooled endpoint of cardiovascular events that includes myocardial infarction (MI), coronary revascularization, congestive heart failure (CHF), or CV mortality. We expect that increased bFGF may itself be a robust marker for increased CV risk in diabetes mellitus for three reasons. First, because bFGF was independently associated with (micro)-albuminuria in type 2 diabetes mellitus. Second, because increased bFGF was associated with increased activity in the renin-angiotensin system in vascular smooth muscle cells (Dzau, et al. JCI, 1995). And third, because (as we reported) angiotensin converting enzyme inhibitor (ACEi) drugs substantially decreased plasma bFGF levels in (micro)- albuminuric diabetes mellitus type 2, and (as others reported) ACEi drugs substantially reduced the risk of development of CHF in patients with LVH 2, the risk of mortality after MI (8,9), and the risk of CV death in diabetic patients with proteinuria.

Because plasma endothelial cell (bFGF) activity correlated significantly with glycemic levels in diabetes mellitus type 2, plasma bFGF may be one of the pathogenetic links between glycemic levels and an increased risk of cardiovascular events in diabetes mellitus, type 2.

Methods: Blood (3 mL EDTA plasma) will be collected from each subject in Years 1, and 2 of the Study at each of 6 local participating VA substudy sites. Because plasma endothelial cell (bFGF-like) bioactivity and bFGFR-IR in vivo are stable for months and years based on our prior published studies (1-3), we anticipate that obtaining 2 specimens, 1 each in Years 1, 2 of the study, will provide sufficient data to model proportional risk.

Results: One hundred and five first cardiovascular events occurred in these 399 subjects.

The best fit model of risk factors associated with the time to first CVD occurrence (in the study) over a seven and one-half year period had as significant predictors: prior cardiovascular event [hazard ratio (HR) 3.378; 95% confidence intervals (CI) 3.079-3.807; P <0.0001), baseline plasma bFGF (HR 1.008; 95% CI 1.002-1.014; P D0.01), age (HR 1.027; 95% CI 1.004-1.051; P D0.019), baseline plasma triglycerides (HR 1.001; 95% CI 1.000-1.002; P D0.02), and diabetes duration-treatment interaction (P D0.03). Intensive glucose-lowering was associated with significantly decreased hazard ratios for CVD occurrence (0.38-0.63) in patients with known diabetes duration of 0-10 years, and nonsignificantly increased hazard ratios for CVD occurrence (0.82-1.78) in patients with longer diabetes duration. Conclusion: High level of plasma bFGF is a predictive biomarker of future CVD occurrence in this population of adult type 2 diabetes.

In conclusion, the present findings suggest that baseline plasma bFGF may be a marker of CVD risk in adult male veterans with type2 diabetes. These results suggest that increased plasma bFGF drive cell proliferation and be involved in the mechanism for increased CVD occurrence in older adults with advanced type2 diabetes mellitus.

Main Manuscript: Basic fibroblast growth factor predicts cardiovascular disease occurrence in participants from the veterans affairs diabetes trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 DM who are no longer responsive to maximum dose of one or more oral agents.

Exclusion Criteria:

* Not a part of the VADT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2@.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are cardiovascular morbidity and mortality. | End of study.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Abraira, MD, Study Chair — Miami VA Healthcare System, Miami, FL
Locations (7):
- United States (7):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - VA Medical Center, Long Beach, Long Beach, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Result] Zimering MB, Anderson RJ, Ge L, Moritz TE; Investigators for the VADT. Increased plasma basic fibroblast growth factor is associated with coronary heart disease in adult type 2 diabetes mellitus. Metabolism. 2011 Feb;60(2):284-91. doi: 10.1016/j.metabol.2010.02.003. Epub 2010 Mar 6. PMID 20206949
- [Result] Zimering MB, Anderson RJ, Moritz TE, Ge L; Investigators for the VADT. Endothelial cell inhibitory autoantibodies are associated with laser photocoagulation in adults from the Veterans Affairs Diabetes Trial. Metabolism. 2009 Jun;58(6):882-7. doi: 10.1016/j.metabol.2009.02.023. PMID 19375761
- [Result] Zimering MB, Anderson RJ, Moritz TE, Ge L; Investigators for the VADT. Low plasma basic fibroblast growth factor is associated with laser photocoagulation treatment in adult type 2 diabetes mellitus from the Veterans Affairs Diabetes Trial. Metabolism. 2009 Mar;58(3):393-400. doi: 10.1016/j.metabol.2008.10.014. PMID 19217457
- [Result] Zimering MB, Anderson RJ, Luo P, Moritz TE; Investigators for the Veterans Affairs Diabetes Trial. Plasma basic fibroblast growth factor is correlated with plasminogen activator inhibitor-1 concentration in adults from the Veterans Affairs Diabetes Trial. Metabolism. 2008 Nov;57(11):1563-9. doi: 10.1016/j.metabol.2008.06.012. PMID 18940395
- [Result] Zimering MB, Pan Z. Autoantibodies in type 2 diabetes induce stress fiber formation and apoptosis in endothelial cells. J Clin Endocrinol Metab. 2009 Jun;94(6):2171-7. doi: 10.1210/jc.2008-2354. Epub 2009 Mar 17. PMID 19293267
- [Result] Zimering MB, Moritz TE, Donnelly RJ. Anti-neurotrophic effects from autoantibodies in adult diabetes having primary open angle glaucoma or dementia. Front Endocrinol (Lausanne). 2013 May 15;4:58. doi: 10.3389/fendo.2013.00058. eCollection 2013. PMID 23720653
- [Result] Zimering MB, Anderson RJ, Ge L, Moritz TE, Duckworth WC; Investigators for the VADT. Basic fibroblast growth factor predicts cardiovascular disease occurrence in participants from the veterans affairs diabetes trial. Front Endocrinol (Lausanne). 2013 Nov 22;4:183. doi: 10.3389/fendo.2013.00183. eCollection 2013. PMID 24319441